CLINICAL TRIAL: NCT02282553
Title: Diagnosis of Upper Gastrointestinal Pathology in Patients With Recurrent/Refractory Iron Deficiency Anaemia: Magnetically Steerable Gastric Capsule Endoscopy Versus Conventional Gastroscopy.
Brief Title: Gastric Capsule Examination for Iron Deficiency Anaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STH18317
Record Dates: First submitted 2014-10-09; First posted 2014-11-04 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetically steerable pill camera (Experimental): Capsule endoscopy uses a swallowable pill camera which passes through the GI tract by the action of peristalsis. The procedure utilizes a battery powered wireless capsule to transmit images of the gastrointestinal tract as it passes through the small intestine. The images are later downloaded to a computer and reviewed by a trained physician. Magnetically steerable gastric capsule endoscopy uses a pill camera containing a small amount of magnetic material, that can be manoeuvred in the gut and intestine by the physician using a handheld magnet. This technique will be compared to conventional gastroscopy which uses a flexible endoscope. Both techniques will be used to diagnose upper gastrointestinal pathology in patients with recurrent/refractory iron deficient anemia.
  Interventions: Device: Magnetically steerable pill camera (Microcam Navi, Intromedic Ltd, Seoul, Korea); Device: Flexible endoscope

INTERVENTIONS:
Device: Magnetically steerable pill camera (Microcam Navi, Intromedic Ltd, Seoul, Korea) — Capsule endoscopy uses a swallowable pill camera which passes through the GI tract by the action of peristalsis. The procedure utilizes a battery powered wireless capsule to transmit images of the gastrointestinal tract as it passes through the small intestine. The images are later downloaded to a computer and reviewed by a trained physician. Magnetically steerable gastric capsule endoscopy uses a pill camera containing a small amount of magnetic material, that can be manoeuvred in the gut and intestine by the physician using a handheld magnet.
Device: Flexible endoscope — The current standard for investigation of upper gastrointestinal disorders is flexible endoscopy; oesophagogastroduodenoscopy (OGD), also known as gastroscopy.
  Other Names: Oesophagogastroduodenoscope

SUMMARY:
This is a pilot prospective single blind controlled trial comparing magnetically steerable gastric capsule endoscopy to conventional oesophagogastroduodenoscopy in diagnosing upper gastrointestinal pathology in patients with recurrent/refractory iron-deficient anaemia.

DETAILED DESCRIPTION:
Gastroscopy (OGD) is a useful test for investigating a variety of suspected upper GI disorders. But it is uncomfortable for patients and incurs the risk of intubation and sedation, plus a large proportion of procedures reveal insignificant or no pathology. Capsule endoscopy (CE) is the investigation of choice for diseases of the small bowel. It is safe, noninvasive and well tolerated.

The use of CE is traditionally restricted to the small bowel, although newer capsules to image the oesophagus and colon are currently in use. Previous capsules have failed to adequately image the stomach due to its large volume and rugal folds. Recently a magnetic capsule and handheld magnet has been developed (Microcam Navi, Intromedic Ltd, Seoul, Korea) to enable an element of manoeuvrability of the capsule. This is unnecessary in the small bowel where the capsule is propelled along its' tubular structure by peristalsis, but in the capacious stomach this may allow the capsule to be steered to examine all areas of the stomach.

The investigators have already conducted two feasibility studies in porcine models with promising results and a trial is currently underway using this equipment to steer the small bowel capsule through the stomach into the duodenum. The next logical step is to compare this technique to the conventional standard of upper GI investigation; OGD. Patients with recurrent or refractory iron deficiency anaemia require a combination of gastroscopy and small bowel capsule endoscopy as part of their diagnostic investigations. The investigators wish to undertake a pilot prospective single blind controlled trial comparing magnetically steerable gastric capsule examination to conventional OGD in diagnosing upper gastrointestinal pathology in patients with recurrent/refractory iron deficiency anaemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years and over.
* Patients with recurrent/refractory iron deficiency anaemia who require a gastroscopy and small bowel capsule endoscopy as part of their diagnostic investigations.

Exclusion Criteria:

* Patients under the age of 20 years.
* Patients with a permanent pacemaker, implantable cardioverter defibrillator or REVEAL device.
* Patients with any electronic/magnetic/mechanically controlled devices e.g. sacral nerve stimulators, bladder stimulators.
* Patients that are pregnant.
* Patients who are unable to understand or speak English.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09-25 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield (pathology reporting form) | Baseline
  As completed on pathology reporting form
Gastric mucosal visibility (Assessed on a 1-5 scale ) | Baseline
  Assessed on a 1-5 scale at specific gastric locations
Patient comfort score (visual analogue and numeric rating scales on Patient Comfort Questionnaire document) | Baseline
  Assessed using visual analogue and numeric rating scales on Patient Comfort Questionnaire document

CONTACTS AND LOCATIONS:
Overall Officials: Mark McAlindon, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Royal Hallamshire Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom